CLINICAL TRIAL: NCT07368465
Title: Determinant Factors in Excessive Gestational Weight Gain: Physical Activity, Nutritional Status, and Anxiety
Status: Recruiting | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025/493
Record Dates: First submitted 2026-01-13; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy; Excessive Gestational Weight Gain
Keywords: physical activity; nutritional status; anxiety
MeSH Terms: conditions — Motor Activity; Anxiety Disorders | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Excessive GWG: Participants will be assessed once in the third trimester and categorized into excessive and non-excessive gestational weight gain groups based on IOM recommendations. Physical activity, dietary intake, and pregnancy-related anxiety will be assessed concurrently.
  Interventions: Other: None (Observational Study)

INTERVENTIONS:
Other: None (Observational Study) — This is an observational study. No intervention is assigned to participants. All assessments are conducted as part of routine data collection without any experimental or behavioral intervention.

SUMMARY:
This study aims to identify which of the following factors-physical activity level, nutritional status, or pregnancy-related anxiety-has the strongest influence on excessive gestational weight gain. Pregnant women in their third trimester who are being followed at Gebze Fatih State Hospital and meet the inclusion criteria will be referred to the Exercise Therapy Laboratory of the Department of Physiotherapy and Rehabilitation, Faculty of Health Sciences, Bezmialem Vakıf University. After being informed about the study and providing written informed consent, participants will undergo a face-to-face assessment. Data will be collected prospectively using a demographic information form, the Pregnancy Physical Activity Questionnaire (PPAQ), a nutritional status assessment form, and a pregnancy-related anxiety questionnaire.

DETAILED DESCRIPTION:
Excessive gestational weight gain is a significant public health concern due to its association with adverse maternal and neonatal outcomes. Multiple factors, including lifestyle behaviors and psychological status, may contribute to excessive weight gain during pregnancy. However, the relative contribution of physical activity, nutritional status, and pregnancy-related anxiety remains unclear.

The primary objective of this prospective observational study is to comprehensively determine which of these variables-physical activity level, nutritional status, or pregnancy-related anxiety-has the most significant effect on excessive gestational weight gain.

The study population will consist of pregnant women in their third trimester who are being followed with a diagnosis of pregnancy at Gebze Fatih State Hospital and who meet the predefined inclusion criteria. Eligible participants will be referred to the Exercise Therapy Laboratory of the Department of Physiotherapy and Rehabilitation, Faculty of Health Sciences, Bezmialem Vakıf University.

After receiving detailed verbal and written information about the study, all participants will be asked to provide written informed consent prior to enrollment. Data collection will be conducted prospectively through face-to-face interviews.

Participants will complete the following assessment tools:

A demographic characteristics form, The Pregnancy Physical Activity Questionnaire (PPAQ) to assess physical activity levels, A nutritional status assessment form to evaluate dietary habits, A pregnancy-related anxiety questionnaire to assess anxiety levels associated with pregnancy.

The collected data will be analyzed to determine the relative impact of physical activity, nutritional status, and pregnancy-related anxiety on excessive gestational weight gain.

ELIGIBILITY:
Inclusion Criteria:

* Being in the 3rd trimester of pregnancy
* Being between 18 and 45 years old
* Having the intellectual capacity to understand and respond to what is read.

Exclusion Criteria:

* High-risk pregnancy
* Multiple pregnancy
* Having a chronic disease such as a systemic, neurological, orthopedic, etc.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only women who are able to conceive are included in our study.
Study Population: Pregnant women in the third trimester attending antenatal care clinics will be evaluated once and classified according to IOM-based gestational weight gain categories.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-01-02 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Excessive Gestational Weight Gain | Single assessment during the third trimester (28-40 weeks of gestation)
  Gestational weight gain classified as excessive or non-excessive according to the Institute of Medicine (IOM) recommendations adjusted for pre-pregnancy body mass index.

SECONDARY OUTCOMES:
Physical Activity Level (MET-hours per week) | Single assessment during the third trimester (28-40 weeks of gestation)
  hysical activity is assessed using the Pregnancy Physical Activity Questionnaire (PPAQ). The questionnaire includes 32 items covering household/care activities, occupational activities, and sports/exercise. Time spent in each activity is multiplied by standardized metabolic equivalent (MET) values to calculate energy expenditure, expressed as MET-hours per week (MET-h/week). Activities are classified by intensity as sedentary (<1.5 METs), light (1.5-3.0 METs), moderate (3.0-6.0 METs), or vigorous (>6.0 METs). Higher MET-hours per week indicate higher levels of physical activity (better outcome).
Daily Energy Intake (kcal/day) | Single assessment during the third trimester (28-40 weeks of gestation)
  Dietary intake is assessed using a 24-hour dietary recall form. Total daily energy intake is calculated in kilocalories per day (kcal/day). Higher values indicate higher daily energy intake.
Pregnancy-Related Anxiety Score | Single assessment during the third trimester (28-40 weeks of gestation)
  Pregnancy-related anxiety is assessed using the Pregnancy-Related Anxiety Scale. The scale consists of 33 items rated on a 4-point Likert scale and includes 9 subscales. Eleven items are reverse-coded. Total scores range from 33 to 132, with higher scores indicating higher levels of pregnancy-related anxiety (worse outcome). The scale has no established cut-off value and can be applied to both primiparous and multiparous pregnant women.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided